CLINICAL TRIAL: NCT02925897
Title: Enhancing Self-care Through Opportunistic Motivational Techniques, Used by Community Nurses, While Caring for Housebound Patients With Long-term Conditions: a Mixed Methods Feasibility Study
Brief Title: Enhancing Self-care in the Housebound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-047
Record Dates: First submitted 2016-09-12; First posted 2016-10-06 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2017-02

CONDITIONS: Chronic Illness
MeSH Terms: conditions — Chronic Disease | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): participants will receive their usual treatment from nurses who have had some training in behaviour change and motivational interviewing.
  Interventions: Behavioral: Behaviour change and motivational interviewing
- Control (No Intervention): The participants will receive their usual treatment from nurses who have had no additional training in behaviour change and motivational interviewing.

INTERVENTIONS:
Behavioral: Behaviour change and motivational interviewing — nurses will help patients to identify health behaviours that they would like to change and to explore their motivation and strengths to achieve this.
  Arms: Intervention

SUMMARY:
The prevalence of people living with problems due to a long-term condition (LTC) such as heart disease, diabetes or arthritis in England exceeds 15 million, and the number of those with more than one LTC continues to grow (LTCs). This population consumes a large proportion of health service resources. Advancing age and LTCs increase the likelihood of becoming housebound, this has a detrimental effect on health and quality of life. Health policy advocates a health service model of empowerment and self-care. People who live with LTCs are often very knowledgeable about how to look after their health but find it difficult to adjust their.

Motivational techniques have been demonstrated to facilitate behaviour change through changing the style of communication from directive to collaborative. The use of patient-centred conversational style of communication has been shown to elicit more willingness to change than professional-led directive consultations. Community nurses are in a unique position to influence housebound patients to play a greater part in caring for themselves, preventing complications in their long-term conditions and further ill health.

This study intends to test the feasibility and acceptability of training community nurses in Understanding Behaviour Change, a communication technique which uses motivational interviewing to guide patients to change their behaviour. The opportunistic use of motivational techniques to create participatory relationships between patients, community nurses potentially represents an effective intervention to enable patients with LTCs to optimise the way they care for themselves.

Motivational interviewing techniques have been widely demonstrated to bring about behaviour change but have not been studied in the context of changing the style of communication between housebound patients and the professionals caring for them.

DETAILED DESCRIPTION:
Study Design and Methods This study has a pragmatic mixed methods explanatory design, consisting of a clinical trial and a qualitative study. The results of the trial will be used to inform the interview protocol for the qualitative study, the data from which will be analysed to explore and elaborate on the results from the trial.

Phase one: Clinical Trial Design This is a parallel controlled, single blinded trial. The outcomes of the patients cared for by nurses who have undergone UBC will be compared with the outcomes from patients who have received usual care.

Population: All patients referred to the caseload of the community nursing teams will be considered for inclusion in this trial. If the patients are on the community caseload they will be considered housebound at the time of treatment as this is the criteria for acceptance onto the caseload. The criteria of infrequent absences from home which are short in duration and require taxing effort is used in line with the Medicare definition of homebound (U.S. Department of Health and Human Services 2010).

Blinding: The patients will not be told whether or not they are being cared for by nurses who have received UBC training.

Randomisation: It is intended that a trial resulting from this study would have a random controlled cluster design to overcome this. All eligible patients in one locality will be exposed to the intervention and all eligible patients in the other locality will not be exposed. Randomising at community nursing team level in a cluster trial could lead to contamination, as within the locality nurses may cover for other teams at weekends and during periods of staff absence. If this feasibility study leads to a larger trial, it would be possible to randomise at locality level to reduce bias. Non-randomised feasibility studies do not have reduced validity (Craig et al 2008).

Setting: This feasibility study is planned to take place within two neighbouring Clinical Commissioning Groups (CCG) that serve a population of 335,000 people (Office for National Statistics 2011). The intervention locality has nine community nursing teams linked to GP practices and grouped as three clusters. The patients in the usual care arm of the trial will be recruited from a neighbouring CCG which has a similar configuration of community nursing teams, including community matrons and specialist nurses. All the nursing working with patients in the intervention cluster will be trained in UBC.

Sample: All patients are potential participants if they are admitted to community caseloads. In the locality where UBC is to be used, all the patients seen by the nurses will be exposed to motivational techniques. The participants will be those patients who are newly and consecutively referred to the caseload of either the intervention community nurse teams or the control teams and are expected to have three or more contacts with the community nurses.

Recruitment procedure All patients are potential participants if they meet the inclusion criteria. Once identified the staff caring for them will explain the study and give them the information sheet. If they are interested in participating they will be given a consent form. They will be contacted the next day by phone to ask if they are willing to participate. If they are willing, at the next visit, the usual carer or the investigator will discuss the study with them and determine their understanding of participating. If they understand they will be asked to sign a consent form. Their part in the trial will consist of completing questionnaires at the start and 3 months into their treatment. The questionnaires will be administered by either a member of the care team or the researcher. The final Questionnaire will be given to them by a member of the usual care team or the researcher. The questionnaires can be administered either face to face or by phone depending on the participants' wishes. Questionnaires will be supplied with envelopes to encourage candid responses. Health service use will be measured through the investigator accessing this data from electronic records, with the patients consent, at referral and three months after intervention.

Intervention: Understanding Behaviour Change (UBC) training. UBC training is structured on the Prevention and Lifestyle Behaviour Change: Competency Framework (National Institute for Health and Clinical Excellence 2007). The training is accredited by the Royal Society for Public Health (RSPB). The training aims to enable learners to understand behaviours associated with active listening, effective hearing, reflecting, checking understanding and their use in effective communication. UBC training also identifies enabling approaches to building relationships, knowledge of behaviour change models and how to explore an individual's motivation to adopt positive health behaviours. The training will enhance the trainees' skills in supporting individuals to develop strategies to enable them to plan and implement changes in their lifestyle or health behaviour. The training is supported with role play to develop communication skills.

Sixteen members of staff from the community nursing team leads, community matrons, and specialist nurses will be trained as motivational champions with UBC consisting of two days of face-to-face training. The motivational Champions will take a multiple-choice exam set by an external examiner to assess their knowledge. The remaining 20 staff will have one session of four hours training, face-to-face, and including role play. The training will be provided by the KCHT Improvement Team in a venue within the locality. The champions will provide supervision and encouragement in the use of the UBC Intervention through monthly action learning sets. The action learning sets will be attended by two motivational champions and two or three other staff. This allows the staff to reflect on their experiences of using UBC and share the learning they have acquired. To evaluate their professional development the champions will be asked to complete a questionnaire before undertaking the training and one month afterwards. This will explore their knowledge and confidence in behaviour change and the barriers and facilitators to implementing their learning. Themes from the questionnaires will be discussed in the action learning sets.

Intervention fidelity All staff will have an assessment of a patient audiotaped and assessed by the researcher for use of UBC using the Peer Proficiency Assessment (PEPA) (Mastroleo et al 2009). This process will be explained to patients when they first consent to being part of the study and again before the recording takes place. The audio-recorder will be encrypted and the recordings will be analysed using the PEPA tool, by the investigator, and then deleted. The PEPA tool was developed to evaluate the fidelity to use of MI skills in undergraduate peer counsellors. PEPA is a valid tool which is simple to use and demonstrates high inter-rater reliability between master coders, experienced peer counsellors and minimally trained peer counsellors (Mastroleo et al 2009).

Phase two: Interview study Aim: To explore the intervention arm patients' experience of the service they receive, their interactions with the nurses and any impact it has on their ability to care for themselves.

Design: Qualitative Method: An interview protocol will be developed, informed by the analysis of the quantitative data. Interviews allow rich data to be collected, guided by topic headings in the specific research area. This creates flexibility and focus but depends upon the interviewer having the skills to listen actively, reflectively and attentively while guiding and controlling the quality of the data (Polit & Beck 2008). Each interview is expected to take about an hour but may be shorter, depending on the wishes and health of the individual patient. The interviews will be audio taped with permission and the interviewer will take additional anonymised notes identifying patients with a unique number.

Sample: Six patients from the intervention group will be interviewed for rich qualitative data, to explore their views and perception of how the community nurses talked to them and any impact it has had on how they care for themselves. The sample to be interviewed will be selected to represent the extremes of results from the Consultation and relational empathy measure (Mercer et al 2004). It is initially intended to interview six participants, but if important themes and differences are found it may be necessary to widen this inquiry to explore the phenomena fully (Kelly 2010).

Analysis: The audiotapes will be transcribed verbatim, by the investigator or an agency used for medical transcription by KCHT, and checked for accuracy by the interviewer. The transcripts will be shared with the patient to check that they are a true representation of their intended meaning. The audio tapes will be deleted after transcription; transcripts will be anonymised using a patient identification number. The transcripts will be read with the notes taken during the interview for meaning. They will be re-read to identify themes that best capture the essential qualities of that interview. Themes from within each section of the transcript will be identified, and possible or likely connections between themes sought. A qualitative code book will be developed. The data will be coded and the codes assigned labels. The codes will be grouped into themes, interrelated and assigned to a smaller set of categories. Computer assisted data analysis software NVivo will be used to organise and support rigorous data analysis (St John & Johnson 2004).

Bias: The researcher, who will not be delivering care to this group of patients, will interview the participants using critical reflexivity, to guard against personal bias, and the writing of memos to acknowledge personal preferences, theoretical leanings and investment in the research process (Polit & Beck 2008).

Integration of quantitative and qualitative results:

The quantitative data will be examined with the data from the qualitative phase, to test and refine the explanations for the outcomes (Cresswell & Plano Clark 2012) and inform the design of a future study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give informed consent
* Patients on the community nurses caseload
* Patients with long-term conditions

Exclusion Criteria:

* Any inclusion criteria not met
* Patients who are not expected to be seen more than three times
* Less than 18 years old.
* Patients who are unable to complete the questionnaire in English.
* Patients who through physical or psychological conditions do not have the potential to contribute to their own care, as decided by the community nurse.
* Patients who are unable to give informed consent.
* Those who hold their own health budget or are part of the proactive care programme
* Patients who are at the end of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention to the study | 12 months
  To test the feasibility of recruiting people who are housebound to a behaviour change
  intervention (ESC) The number of housebound patients who meet the inclusion criteria of those who is recruited to the study.
  The number of participants who complete the study. The reasons for not completing the study.

SECONDARY OUTCOMES:
The appropriateness of the preliminary primary outcome | 12 months
  Patient centeredness to be collected at three months (T2) using the Consultation and relational empathy measure. This is a 10 item questionnaire with a 5 point Likert Scale 0=poor to 5=excellent.
Measurement of patient enablement | 12 months
  Patient enablement tool:This is a six-question instrument each of which have four possible response options much better, better, worse or the same or not applicable
General self-efficacy scale | 12 months
  This is a 12 item Likert scale which is used to assess patients' confidence in their ability to change health behaviours and achieve goals
Quality of life | 12 months
  EQ-5D which measures five dimensions of health: mobility, self-care, ability to carry out usual activities, pain or discomfort and anxiety and depression. These dimensions are each scored on five levels.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley R Sage, Principal Investigator — King's College London
Locations (1):
- Kent Community Health Foundation Trust, Maidstone, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no individual participant data will be made available